CLINICAL TRIAL: NCT07171242
Title: Shanghai Prospective Registry Study of Ischemic Stroke
Acronym: 4S
Status: Recruiting | Type: Observational
Sponsor: Qiang Dong (Other)
Responsible Party: Sponsor-Investigator, Qiang Dong, Director, Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: KY2024-1385
Record Dates: First submitted 2025-08-25; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute ischemic stroke group: Collect basic clinical information about patients, including age, gender, medical history, etc.

SUMMARY:
This study aims to conduct a prospective cohort study on patients with imaging-confirmed ischemic stroke based on the 4S database. The primary objectives are to investigate the incidence, clinical characteristics, risk factors, and pathophysiological mechanisms of young-onset stroke, as well as to analyze the evolving trends in the etiology of young-onset stroke in the Shanghai region over recent years. This includes examining the roles of traditional risk factors (such as hypertension and diabetes) and emerging factors (such as air pollution and lifestyle changes), and exploring the associations between these factors and patient outcomes. Additionally, the study will analyze the association between reperfusion therapies such as intravenous thrombolysis, acute-phase management, and secondary prevention with clinical outcomes. Finally, it will delve into the screening, treatment, and challenges associated with genetic young stroke patients with Farby syndrome, providing comprehensive information for regional stroke prevention and control strategies targeting young stroke patients.

DETAILED DESCRIPTION:
This study is designed as a prospective cohort investigation utilizing data from the 4S database, focusing specifically on patients with imaging-confirmed ischemic stroke who are classified as having young-onset stroke (typically defined as occurring in individuals under 55 years of age). The purpose is to provide a thorough understanding of stroke in younger populations within the Shanghai region through collecting relevant clinical information of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older diagnosed with acute or subacute ischemic stroke
2. The diagnosis of stroke must be confirmed through clinical assessment and imaging examinations
3. In cases where imaging examinations are negative or unavailable, the clinical diagnosis of stroke must be confirmed by an experienced neurologist. (4)Patients must sign an informed consent form agreeing to the collection of information.

Exclusion Criteria:

1. The amount of missing data exceeds 40% of the data to be entered;
2. After enrollment, it is discovered that the study participant does not meet the inclusion criteria or meets any of the exclusion criteria;
3. Missing persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older diagnosed with acute or subacute ischemic stroke
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient general information | Upon admission
  Name, age, gender, place of residence, date of admission, name of hospital, hospital grade, TOAST classification
Risk factors (assessed by medical history review and clinical evaluation) | Upon admission
  The presence (Yes) or absence (No) of each listed risk factor will be determined for each participant through medical history review and clinical evaluation：Smoking, hypertension, atrial fibrillation, hyperlipidemia, diabetes, history of cerebral infarction, myocardial infarction, other heart diseases, dementia, chronic obstructive pulmonary disease, history of bleeding or bleeding tendency
Pre-illness medication history（assessed by medical history review） | Upon admission
  The use of the following pre-illness medication categories, as confirmed by medical history review upon admission, will be recorded as a binary outcome (Yes/No) for each participant: antihypertensive drugs, antidiabetic drugs, lipid-lowering drugs, anticoagulants, antiplatelet drugs.
Baseline National Institutes of Health Stroke Scale (NIHSS) Score | Upon admission
  The severity of neurological deficit will be assessed using the National Institutes of Health Stroke Scale (NIHSS) upon admission. The NIHSS is a 15-item neurologic examination stroke scale with scores ranging from 0 to 42, where higher scores indicate more severe neurological deficit.
Pre-Stroke Modified Rankin Scale (mRS) Score | Prior to stroke admission (assessed upon current admission)
  Functional ability prior to stroke admission will be assessed using the Modified Rankin Scale (mRS). The mRS is a 6-point disability scale ranging from 0 (no symptoms) to 5 (severe disability), with a separate score of 6 indicating death. Higher scores indicate worse functional outcome.
Time Metrics from Symptom Onset to Hospital Presentation | Upon admission
  The following time points will be recorded to determine delays in presentation: time when the patient was last known to be at their normal neurological baseline, time of symptom onset, and time of arrival at the hospital.
Number of Participants Undergoing Reperfusion Therapy | Within 24 hours of admission
  The administration of specific reperfusion therapies during hospitalization will be recorded as a binary outcome (Yes/No) for each participant. Therapies include: intravenous thrombolysis and endovascular treatment (mechanical thrombectomy). Determination will be made through review of medical records and procedure documentation.
Number of Participants With Baseline Neuroimaging Findings | At admission (within 24 hours of hospitalization)
  The presence of findings on baseline neuroimaging (CT or MRI) performed at admission will be recorded. This includes the presence of cerebral small vessel disease manifestations (e.g., white matter hyperintensities, lacunes) and the location and degree of large vessel occlusion/stenosis.
Number of Participants With Cardiac Evaluation Findings | Within 7 days of admission
  Results from cardiac evaluations performed during hospitalization will be recorded as binary outcomes (normal/abnormal). Assessments include: echocardiogram (cardiac ultrasound), electrocardiogram (ECG), 24-hour Holter monitoring, and bubble test (for patent foramen ovale detection).
Modified Rankin Scale (mRS) Score at Discharge | Day 7 post-stroke (or at discharge if earlier)
  Functional outcome at discharge will be assessed using the Modified Rankin Scale (mRS). The mRS is a 7-point disability scale ranging from 0 (no symptoms) to 6 (death), where higher scores indicate worse functional outcome.
Discharge Diagnosis | Day 7 post-stroke (or at discharge if earlier)
  The primary diagnosis documented in the medical record at the time of hospital discharge will be recorded.
Length of Hospital Stay | Up to 30 days (from admission to discharge，this will be calculated from admission to discharge for each participant)
  The duration of hospitalization, calculated as the number of days from admission to discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yaghi S, Henninger N, Giles JA, Leon Guerrero C, Mistry E, Liberman AL, Asad D, Liu A, Nagy M, Kaushal A, Azher I, Mac Grory B, Fakhri H, Brown Espaillat K, Pasupuleti H, Martin H, Tan J, Veerasamy M, Esenwa C, Cheng N, Moncrieffe K, Moeini-Naghani I, Siddu M, Scher E, Trivedi T, Furie KL, Keyrouz SG, Nouh A, de Havenon A, Khan M, Smith EE, Gurol ME. Ischaemic stroke on anticoagulation therapy and early recurrence in acute cardioembolic stroke: the IAC study. J Neurol Neurosurg Psychiatry. 2021 Oct;92(10):1062-1067. doi: 10.1136/jnnp-2021-326166. Epub 2021 Apr 26. PMID 33903185
- [Result] Brouwer J, Smaal JA, Emmer BJ, de Ridder IR, van den Wijngaard IR, de Leeuw FE, Hofmeijer J, van Zwam WH, Martens JM, Roos YBWEM, Majoie CB, van Oostenbrugge RJ, Coutinho JM; MR CLEAN Registry Investigatorsdagger. Endovascular Thrombectomy in Young Patients With Stroke: A MR CLEAN Registry Study. Stroke. 2022 Jan;53(1):34-42. doi: 10.1161/STROKEAHA.120.034033. Epub 2021 Dec 7. PMID 34872339
- [Result] Shu L, Akpokiere F, Mandel DM, Field TS, Leon Guerrero CR, Henninger N, Muppa J, Affan M, Haq Lodhi OU, Heldner MR, Antonenko K, Seiffge DJ, Arnold M, Salehi Omran S, Crandall R, Lester E, Lopez-Mena D, Arauz A, Nehme A, Boulanger M, Touze E, Sousa JA, Sargento-Freitas J, Barata V, Castro-Chaves P, Brito MT, Khan M, Mallick D, Rothstein A, Khazaal O, Kaufmann JE, Engelter ST, Traenka C, Aguiar de Sousa D, Soares MD, Rosa SB, Zhou L, Gandhi P, Mancini S, Metanis I, Leker RR, Pan K, Dantu V, Baumgartner K, Burton TM, Von Rennenberg R, Nolte CH, Choi R, MacDonald J, Bavarsad Shahripour R, Guo X, Ghannam M, Almajali M, Samaniego EA, Rioux B, Zine-Eddine F, Poppe A, Fonseca AC, Baptista MF, Cruz D, Romoli M, De Marco G, Longoni M, Keser Z, Griffin KJ, Kuohn L, Frontera JA, Amar JY, Giles JA, Zedde M, Pascarella R, Grisendi I, Nzwalo H, Liebeskind DS, Molaie A, Cavalier A, Kam W, Mac Grory B, Al Kasab S, Anadani M, Kicielinski KP, Eltatawy A, Chervak L, Chulluncuy Rivas R, Aziz YN, Mistry EA, Bakradze E, Tran TL, Rodrigo-Gisbert M, Requena M, Saleh Velez FG, Garcia JO, Muddasani V, de Havenon A, Sanchez S, Vishnu VY, Yaddanapudi S, Adams L, Browngoehl A, Ranasinghe T, Dunston R, Lynch Z, Penckofer M, Siegler JE, Mayer S, Willey JZ, Zubair AS, Cheng YK, Sharma R, Marto JP, Krupka D, Klein P, Nguyen TN, Asad SD, Sarwat Z, Balabhadra A, Patel S, Secchi T, Martins SC, Mantovani GP, Kim YD, Krishnaiah B, Elangovan C, Lingam S, Qureshi AY, Fridman S, Alvarado A, Khasiyev F, Linares G, Mannino M, Terruso V, Tountopoulou A, Tentolouris-Piperas V, Martinez-Marino MM, Carrasco Wall V, Indraswari F, El Jamal SE, Liu S, Zhou M, Alvi MM, Ali F, Sarvath M, Morsi RZ, Kass-Hout T, Shi F, Zhang J, Sokhi D, Said J, Mongare N, Simpkins AN, Gomez R, Sen S, Ghani M, Elnazeir M, Wangqin R, Xiao H, Kala NS, Khan F, Stretz C, Mohammadzadeh N, Goldstein ED, Furie K, Yaghi S. Intravenous Thrombolysis in Patients With Cervical Artery Dissection: A Secondary Analysis of the STOP-CAD Study. Neurology. 2024 Oct 8;103(7):e209843. doi: 10.1212/WNL.0000000000209843. Epub 2024 Sep 19. PMID 39298709
- [Result] Verhoeven JI, van Lith TJ, Ekker MS, Hilkens NA, Maaijwee NAM, Rutten-Jacobs LCA, Klijn CJM, de Leeuw FE. Long-term Risk of Bleeding and Ischemic Events After Ischemic Stroke or Transient Ischemic Attack in Young Adults. Neurology. 2022 Aug 9;99(6):e549-e559. doi: 10.1212/WNL.0000000000200808. Epub 2022 Jun 2. PMID 35654598
- [Result] Verburgt E, Hilkens NA, Ekker MS, Schellekens MMI, Boot EM, Immens MHM, van Alebeek ME, Brouwers PJAM, Arntz RM, van Dijk GW, Gons RAR, van Uden IWM, den Heijer T, van Tuijl JH, de Laat KF, van Norden AGW, Vermeer SE, van Zagten MSG, van Oostenbrugge RJ, Wermer MJH, Nederkoorn PJ, Kerkhoff H, Rooyer FA, van Rooij FG, van den Wijngaard IR, Ten Cate TJF, Tuladhar AM, de Leeuw FE, Verhoeven JI. Short-Term and Long-Term Risk of Recurrent Vascular Event by Cause After Ischemic Stroke in Young Adults. JAMA Netw Open. 2024 Feb 5;7(2):e240054. doi: 10.1001/jamanetworkopen.2024.0054. PMID 38376841
- [Result] Joglar JA, Chung MK, Armbruster AL, Benjamin EJ, Chyou JY, Cronin EM, Deswal A, Eckhardt LL, Goldberger ZD, Gopinathannair R, Gorenek B, Hess PL, Hlatky M, Hogan G, Ibeh C, Indik JH, Kido K, Kusumoto F, Link MS, Linta KT, Marcus GM, McCarthy PM, Patel N, Patton KK, Perez MV, Piccini JP, Russo AM, Sanders P, Streur MM, Thomas KL, Times S, Tisdale JE, Valente AM, Van Wagoner DR; Peer Review Committee Members. 2023 ACC/AHA/ACCP/HRS Guideline for the Diagnosis and Management of Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2024 Jan 2;149(1):e1-e156. doi: 10.1161/CIR.0000000000001193. Epub 2023 Nov 30. PMID 38033089
- [Result] Ekker MS, Boot EM, Singhal AB, Tan KS, Debette S, Tuladhar AM, de Leeuw FE. Epidemiology, aetiology, and management of ischaemic stroke in young adults. Lancet Neurol. 2018 Sep;17(9):790-801. doi: 10.1016/S1474-4422(18)30233-3. PMID 30129475
- [Result] Bejot Y, Daubail B, Jacquin A, Durier J, Osseby GV, Rouaud O, Giroud M. Trends in the incidence of ischaemic stroke in young adults between 1985 and 2011: the Dijon Stroke Registry. J Neurol Neurosurg Psychiatry. 2014 May;85(5):509-13. doi: 10.1136/jnnp-2013-306203. Epub 2013 Nov 18. PMID 24249786
- [Result] Ekker MS, Verhoeven JI, Vaartjes I, van Nieuwenhuizen KM, Klijn CJM, de Leeuw FE. Stroke incidence in young adults according to age, subtype, sex, and time trends. Neurology. 2019 May 21;92(21):e2444-e2454. doi: 10.1212/WNL.0000000000007533. Epub 2019 Apr 24. PMID 31019103
- [Result] Madsen TE, Khoury JC, Leppert M, Alwell K, Moomaw CJ, Sucharew H, Woo D, Ferioli S, Martini S, Adeoye O, Khatri P, Flaherty M, De Los Rios La Rosa F, Mackey J, Mistry E, Demel SL, Coleman E, Jasne A, Slavin SJ, Walsh K, Star M, Broderick JP, Kissela BM, Kleindorfer DO. Temporal Trends in Stroke Incidence Over Time by Sex and Age in the GCNKSS. Stroke. 2020 Apr;51(4):1070-1076. doi: 10.1161/STROKEAHA.120.028910. Epub 2020 Feb 12. PMID 32078459

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT07171242/Prot_SAP_ICF_000.pdf